CLINICAL TRIAL: NCT05671978
Title: Effect of Head Elevated Position on Ease of Tracheal Intubation Using Hyper-angulated Video-laryngoscope in Patients With Simulated Difficult Airway
Brief Title: Head Elevated Position and Hyper-angulated Video-laryngoscope Guided Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, Associate Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-11-010-001
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neutral position (Placebo Comparator): intubation was performed in the neutral position
  Interventions: Procedure: neutral position
- back-up head elevated position (Experimental): he trachea was intubated in the back-up head elevated position
  Interventions: Procedure: back-up head elevated position

INTERVENTIONS:
Procedure: back-up head elevated position — The patient was then placed in the back-up head elevated position to align the external auditory meatus and sternal notch, which was achieved by breaking the operating table
  Arms: back-up head elevated position
Procedure: neutral position — The patient was then placed in the netural position
  Arms: neutral position

SUMMARY:
Cervical immobilization with manual in-line stabilization (MILS) is recommended to prevent further neurologic injury during intubation in patients with known or suspected cervical spine injuries. However, MILS is associated with increased rates of failed tracheal intubation using direct laryngoscopy, because the restriction of neck flexion and head extension may prevent adequate alignment of the oral, pharyngeal, and tracheal axes, hence adversely affecting laryngeal visualization during direct laryngoscopy.

The GlideScope® (Verathon, Bothell, WA, USA) is a videolaryngoscope with an hyer-angulated blade (HA-VL), which is characterized by a sharper curvature than the Macintosh blade. The large curvature of the HA-VL allows seeing 'round the corner', which can provide indirect laryngeal visualization even with restricted neck movements . However, the HA-VL also prevents direct visualization of larynx, which make it difficult to guide the tracheal tube (TT) towards the glottis despite obtaining a good laryngeal view. Thus, the good view of the laryngeal inlet provided by videolaryngoscopes does not always lead to an easy or successful intubation. There are numerous reports in the literature of devices managing to achieve an improvement in view but still being unable to pass an TT to laryngeal inlet. Thus, the key to a successful tracheal intubation using HA-VL lies not in the laryngeal view obtained but in the ease of inserting the TT. Recent meta studies comparing alternative intubation devices with the standard Macintosh laryngoscope in subjects with cervical spine immobilization reported that GlideScope® was associated with improved glottis visualization but no statistically significant differences in intubation failure or time to intubation compared with direct laryngoscopy.

The sniffing position recommended for direct laryngoscopy has been reported to interfere with successful tracheal intubation with HA-VL because flexion of the neck narrows the angle between the sternum and the chin, making it more difficult to insert the HA-VL blade into mouth. In contrast, placing the patient in a 'neutral' or 'back-up head-elevated (BUHE)' position was not associated with a higher incidence of difficult laryngoscope with HA-VL. Given that the 'BUHE' position, when compared with the regular supine position, extend the safe apnoea time during direct laryngoscopy, this position seems better suited for HA-VL than neutral position. However, there is currently insufficient evidence to recommend a specific patient position for the use of HA-VL.

Previous studies using magnetic resonance imaging (MRI) suggests that head elevation until the external auditory meatus and sternal notch (AM-S) are in the horizonal plane leads to better anatomic alignment of the pharyngeal and laryngeal axes. Investigators therefore hypothesized that BUHE position (to align the AM-S in horizontal plane), compared with neutral position, would allow a relatively straight passage which makes it easier to guide the TT into the laryngeal inlet (facilitates insertion of TT into the laryngeal entrance) during HA-VL guided intubation. To compare the effect of the BUHE position and the neutral position on the ease of tracheal intubation using a HA-VL (GlideScope®), MILS was applied to patients without any known or suspected neck pathology as a way of simulating a difficult airway. The primary outcome was the tracheal intubation time with both positions. Secondary outcomes examined included rates of successful tracheal intubation and intubation success rate, number of intubation attempts, heart rate responses during intubation, and handling of the Glidesope VL after alignment of the EAM and sternal notch.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA physical status 1-2 who were scheduled for elective surgery under general anaesthesia requiring tracheal intubation.

Exclusion Criteria:

* if they required rapid sequence induction;
* history of previous difficult direct laryngoscopy
* unwilling to provide informed consent
* uncontrolled hypertension
* history of ischaemic heart disease without optimal control of symptoms
* history of acute or recent stroke or myocardial infarction
* cervical spine instability or cervical myelopathy
* symptomatic asthma or reactive airway disease requiring daily pharmacological treatment for control of symptoms
* history of gastric reflux.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
ease of tracheal intubation (easy/modified/unachievable) | The time from the insertion of laryngoscope into oral cavity until tracheal intubation over 1minute period
  the need for optimization procedure to facilitate laryngeal visualization and tracheal intubation easy: no need for optimization procedure. modified: need for optimization procedure unachievable: unable to insert tracheal tube even after optimzation procedure

SECONDARY OUTCOMES:
intubation time | : The time from the insertion of laryngoscope into oral cavity until its removal over 1 minute period
  time required for intubation
percentage of glottic opening (POGO) score (0-100%) | During laryngeal visualization by laryngoscope over 1 minute period
  percentage of glottic opening (0 - 100) 0%: visualization of none of the glottis 100%: visualization of the whole glottis

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SH, Kim KM, Choi EM, Son JM, Park J, Jun JH. Effect of head-elevated versus neutral position on tracheal intubation using a hyper-angulated video laryngoscope under cervical spine immobilization: a randomised crossover trial. Anaesth Crit Care Pain Med. 2025 Dec 3:101720. doi: 10.1016/j.accpm.2025.101720. Online ahead of print. PMID 41349843